CLINICAL TRIAL: NCT03005314
Title: Detection of Circulating Tumor Tells as The Guidance of the Neoadjuvant Chemotherapy of Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); Wuhan YZY Medical Science and Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Xiaogang Zhao, vice- director, The Second Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016YFC0106005
Record Dates: First submitted 2016-08-04; First posted 2016-12-29 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer TNM Staging Primary Tumor (T) T3
MeSH Terms: interventions — Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Other): Postoperative chemotherapy group
  Interventions: Procedure: Surgery
- Chemotherapy (Other): Preoperative chemotherapy group
  Interventions: Procedure: chemotherapy

INTERVENTIONS:
Procedure: chemotherapy — chemotherapy before surgery
  Arms: Chemotherapy
Procedure: Surgery — chemotherapy after surgery
  Arms: Surgery

SUMMARY:
Esophageal carcinoma is a common digestive system tumor, with number of deaths ranking No. 4 in malignant tumors. Esophageal squamous cell carcinoma in stage Ⅱ, III is the most common in China. The esophageal cancer during these stages is no longer localized lesions, and cancer will be transferred to other organs of the body through blood transmission, leading to tumor metastasis, which is the main cause of the patients' death. The tumor cells invade the surrounding tissues of primary tumor cells and enter the blood and lymphatic system, thus the circulating tumor cells (CTC) is formed and transported to a distal tissue, then effusing, adapting to the new microenvironment and finally forming metastases through the process of seeding, proliferation and colonization.

Recently, the controversy of surgical treatment of esophageal carcinoma is concentrated on the neoadjuvant therapy during perioperative period. NCCN guideline of 2015 recommended that patients with esophageal squamous cell carcinoma in T1b, N + and T2-T4a, N0-N + may consider preoperative neoadjuvant therapy, but its supporting literature (David Cunningham 2006, Marc Ychou 2011 and P. van Hagen, 2013) includes patients with pathology of the type adenocarcinoma. The esophageal cancer treatment guidelines of Japan 2015 adopted the opinion of NCCN Guidelines, and recommended neoadjuvant chemotherapy and radical surgery as the standard treatment for stage II and III esophageal cancer patients based on the results of randomized controlled clinical trial JCOG9907. However, the guidelines also pointed out that the role of neoadjuvant chemotherapy for resectable T1-3N0-1M0 cancers remains unclear according to the results of some meta-analysis.

The investigators choose the detection of peripheral venous blood CTCs and the disease-free survival as the main index, to compare the treatment effect of patients, those received neoadjuvant therapy, surgery and those received directly surgery, postoperative chemotherapy with esophageal squamous cell carcinoma in stage Ⅱ, III by means of evidence-based medicine; Define the indication of neoadjuvant chemotherapy in the treatment of esophageal squamous cell carcinoma in stage Ⅱ, III; Draft the solution to evaluate the treatment effect of neoadjuvant chemotherapy to esophageal cancer in stage Ⅱ, III, and the indication of neoadjuvant chemotherapy by test the peripheral venous blood CTCs and join the Chinese clinical guideline.

DETAILED DESCRIPTION:
Background Esophageal carcinoma is a common digestive system tumor, with number of deaths ranking No. 4 in malignant tumors. Surgery is the preferred method of treatment for esophageal cancer, but the local recurrence rate is as high as between 40% and 60%, and 5-year overall survival is only about 30%. Most of esophageal cancers are found in the middle and late stage, losing the chance of operation. Esophageal squamous cell carcinoma in stage Ⅱ, III is the most common in China. The esophageal cancer during these stages is no longer localized lesions, and cancer will be transferred to other organs of the body through blood transmission, leading to tumor metastasis, which is the main cause of the patients' death. The tumor cells invade the surrounding tissues of primary tumor cells and enter the blood and lymphatic system, thus the circulating tumor cells (CTC) is formed and transported to a distal tissue, then effusing, adapting to the new microenvironment and finally forming metastases through the process of seeding, proliferation and colonization. In recent years, as liquid pathology, CTCs are used for several studies of tumor, including the auxiliary diagnosis, recurrence and metastasis detection, prognosis, individualized treatment, medical screening, development of new targeted cancer therapy drugs, searching for a new target for cancer therapy, exploring the mechanism of drug resistance, etc.

Recently, the controversy of surgical treatment of esophageal carcinoma is concentrated on the neoadjuvant therapy during perioperative period. Neoadjuvant therapy has been widely studied in recent years. Compared to the postoperative radiochemotherapy,the preoperative chemotherapy is less toxic and better tolerated. Pure radiotherapy could only work on the local tumor, yet without lethal effect towards micrometastases and CTCs. Studies have shown that neoadjuvant radiotherapy can only improve the resection rate, but could not prolong the patient's survival; the advantages of neoadjuvant chemotherapy include: 1. lower tumor stage, reduce tumor volume , and increase the resection rate; 2. control and treat the tiny metastasis, reduce the recurrence rate; 3. chemotherapeutic drugs can reach to tumor issues with sufficient amount , through the undamaged blood supply system; 4. assess the chemosensitivity of drug in body to guide postoperative treatment.

NCCN guideline of 2015 recommended that patients with esophageal squamous cell carcinoma in T1b, N + and T2-T4a, N0-N + may consider preoperative neoadjuvant therapy, but its supporting literature (David Cunningham 2006, Marc Ychou 2011 and P. van Hagen, 2013) includes patients with pathology of the type adenocarcinoma. The esophageal cancer treatment guidelines of Japan 2015 adopted the opinion of NCCN Guidelines, and recommended neoadjuvant chemotherapy and radical surgery as the standard treatment for stage II and III esophageal cancer patients based on the results of randomized controlled clinical trial JCOG9907. However, the guidelines also pointed out that the role of neoadjuvant chemotherapy for resectable T1-3N0-1M0 cancers remains unclear according to the results of some meta-analysis. But at least for the present studies, compared to direct surgery group, the patients received neoadjuvant therapy did not show inferior effect at aspects such as radical surgery, postoperative complications, disease-free survival and overall survival.

The effect and necessity of neoadjuvant chemotherapy to esophageal squamous cell carcinoma patients in stage Ⅱ, Ⅲ, and its influence to disease-free survival still lack authoritative evidence-based medical support, is a clinical urgency need to be solved.

Research objectives Choose the detection of peripheral venous blood CTCs and the disease-free survival as the main index, to compare the treatment effect of patients, those received neoadjuvant therapy, surgery and those received directly surgery, postoperative chemotherapy with esophageal squamous cell carcinoma in stage Ⅱ, III by means of evidence-based medicine; Define the indication of neoadjuvant chemotherapy in the treatment of esophageal squamous cell carcinoma in stage Ⅱ, III; Draft the solution to evaluate the treatment effect of neoadjuvant chemotherapy to esophageal cancer in stage Ⅱ, III, and the indication of neoadjuvant chemotherapy by test the peripheral venous blood CTCs and join the Chinese clinical guideline.

Main research content:

Design dual-center (Second Hospital of Shandong University and Shandong Cancer Hospital Affiliated to Shandong University) prospective clinical contrast trials by selecting the preoperative patients with esophageal squamous cell carcinoma in clinical stage Ⅱ, III. Complete the work of patients screening, informed consent, preoperative preparation, surgery, neoadjuvant chemotherapy and follow-up visits under the guide of Standardized treatment program. Detect the CTCs by extract the peripheral venous blood at the time of the day before initial treatment (neoadjuvant chemotherapy or surgery), one week after surgery and the follow-up visits of 3 months, 6 months, 1 year, 2years after surgery. The main evaluation index of the study is the change of CTCs in peripheral blood and the survival period of disease-free of patients, with secondary evaluation index including the surgery effect, pathology, recurrence rate of the patients, long-term survival as well as other prognostic indicators. Assess the guidance of CTCs detection towards neoadjuvant chemotherapy in the treatment of esophageal squamous carcinoma in stage Ⅱ, III.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven squamous cell carcinoma of the thoracic esophagus;clinical stage II or III excluding T4 disease
* resectable disease; ECOG performance status of 0 to 2
* no previous chemo- or radiotherapy for any malignancies
* sufficient organ function.

Exclusion Criteria:

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
progression- free survival | through study completion, an average of 2-3 year
  survival without recurrence or metastasis

SECONDARY OUTCOMES:
overall survival | through study completion, an average of 5 year
  postoperation to death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Doctor, Principal Investigator — The Second Hospital of Shandong University
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No